CLINICAL TRIAL: NCT02371668
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study in Healthy Volunteers to Evaluate the Efficacy and Safety of CR6261 in an H1N1 Influenza Healthy Human Challenge Model
Brief Title: Efficacy and Safety of CR6261 in an H1N1 Influenza Healthy Volunteer Human Challenge Model
Acronym: CR6261
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 150069; 15-I-0069 (Other: NIAID)
Record Dates: First submitted 2015-02-25; First posted 2015-02-26 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2018-11-30

CONDITIONS: H1N1 Influenza Healthy Volunteers
Keywords: Influenza A; H1N1; Challenge Model; Human Immunoglobulin and H1N1; Efficacy and Safety in H1N1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo, 5% dextrose (D-glucose) water
  Interventions: Biological: Placebo
- CR6261 (Experimental): CR6261, Investigational monoclonal antibody against influenza A viruses
  Interventions: Biological: CR6261

INTERVENTIONS:
Biological: CR6261 — 50 mg/kg administered as a single 2-hour intravenous infusion on Day 1 (24 hours after virus administration).
  Arms: CR6261
Biological: Placebo — Administered as a single 2-hour intravenous infusion on Day 1 (24 hours after virus administration).
  Arms: Placebo

SUMMARY:
Background:

- Researchers want to see if a new drug reduces flu disease in people treated with this drug versus a placebo. The drug has an antibody that may help the immune system fight the flu. Placebo is only sugar and water. All participants will get the flu virus. They may or may not develop flu symptoms.

Objective:

- To see if the drug CR6261 reduces flu disease in people treated with this drug versus a placebo.

Eligibility:

- Healthy nonsmokers ages 18 45.

Design:

* Participants will be screened under a separate protocol.
* Participants must use contraception or abstinence for several weeks before and after the study. They must have no alcohol for 1 day before each visit. Any medicine must be approved by the study doctor until after follow-up.
* Participants will stay in a hospital isolation unit for at least 10 days.
* They will have:
* Medical history
* Physical exam
* Blood and urine tests
* Heart and lung test
* Tests for drugs and alcohol
* Throughout their stay, participants will:
* Be closely watched by a medical team
* Have nasal washes and swabs several times a day
* Participants will have the flu virus sprayed in each nostril.
* The next day, participants will get either study drug or placebo through a soft plastic tube placed in a vein by needle. It will take 2 hours. They will not know which they get.
* Participants can go home after 10 days if they test negative for the flu 2 days in a row.
* Participants will have daily questionnaires at home and 2 follow-up visits over 2 months.

DETAILED DESCRIPTION:
The high morbidity and mortality associated with both pandemic and seasonal influenza and the threat of new potentially pandemic strains emerging makes influenza an important infectious disease and public health problem. Mean annual estimates of influenza deaths due to seasonal influenza alone attributes up to 49,000 deaths in the US and 250,000 to 500,000 deaths in industrialized countries to influenza. Pandemics can have an even more devastating effect. Public health agencies must continue to be prepared by making attempts to reduce the public health impact of this important virus.

In the realm of influenza therapeutics, antiviral drugs are currently used to treat influenza infection in those who fail to be protected by current vaccines or those who do not receive a vaccine. Currently, only two classes of antivirals are FDA approved for the treatment of influenza A: neuraminidase inhibitors and matrix M2 channel blockers. Although these drugs have been shown to be effective in reducing influenza illness by 24-48 hours and reducing shedding in relatively healthy adults, as with vaccination, they have had limited effectiveness in high risk groups and those who have severe or complicated influenza infections. In addition, antiviral resistance has become very common in human influenza A viruses, as currently circulating H1N1 and H3N2 strains are resistant to the adamantane M2 channel blockers and many cases of neuraminidase inhibitor resistance have also been reported with strains of both subtypes. This resistance can develop quickly and in most cases only requires a single amino acid change. Given these significant issues with currently available treatments, novel therapies for influenza are clearly needed.

Live virus challenge studies have played a pivotal role in developing influenza therapeutics in the past, and they will be instrumental in the future. No novel therapeutic or prophylactic agent has been FDA-approved since the last influenza challenge studies ceased over a decade ago. In collaboration with the Crucell Vaccine Institute (part of Crucell which is in the Janssen family of Pharmaceutical Companies of Johnson & Johnson) this protocol will evaluate mAb CR6261 for possible therapeutic value. Unlike the current antivirals that are compounds which interfere with some portion of the viral replicative cycle, this agent is a mAb that targets the stem of HA, neutralizing the virus by stabilizing the pre-fusion state and preventing the pH-dependent fusion of viral and cellular membranes. Pre-clinical data suggest that this mAb has good cross-protective efficacy with a variety of HA subtypes unlike current vaccines, making it potentially effective in the event of an emerging influenza virus outbreak with a novel HA subtype. In addition, the conserved nature of the HA stem region suggests that amino acid changes conferring resistance are much less likely. We will effort to demonstrate that CR6261 leads to improved outcomes compared with placebo with respect to the AUC of virus shedding as determined by qPCR in NP swabs in all treated subjects.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Greater than or equal to 18 and less than or equal to 45 years of age.
2. Non-smoker.
3. Willingness to remain in isolation for the duration of viral shedding (at a minimum 10 days) and to comply with all study requirements.
4. A male subject is eligible for the study if he agrees to practicing abstinence or using a condom with spermicide plus an acceptable form of contraception (see inclusion criteria 5) being used by any female partner from 4 weeks before to 12 weeks after intranasal challenge with influenza.
5. A female participant is eligible for this study if she is not pregnant or breast feeding and 1 of the following:

   * Of nonchildbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses in greater than or equal to 1 year).
   * Of childbearing potential but agrees to practice effective contraception or abstinence for 4 weeks prior to and 8 weeks after administration of the influenza challenge virus. Acceptable methods of contraception include a male partner who is sterile and is the sole sexual partner of the female participant or a male partner who uses a condom with spermicide plus 1 or more of the following: 1) implants of levonorgestrel; 2) injectable progestogen; 3) an intrauterine device with a documented failure rate of <1%; 4) oral contraceptives; and 5) double barrier method including diaphragm.
6. Willing to have samples stored for future research.
7. Prechallenge serum HAI titer against the challenge virus less than or equal to 1:10 within 60 days of admission for the study.
8. HIV uninfected confirmed by testing within 60 days of admission for the study.
9. Agrees to abstain from alcohol intake 24 hours before admission on Day -1, during the inpatient period of the study, and 24 hours prior to all other outpatient clinic visits.
10. Agrees to not use over-the-counter medications (including aspirin, decongestants, antihistamines, and other NSAIDs), and herbal medication (including, but not limited to, herbal tea, St. John s Wort), within 14 days prior to study drug administration through the final follow-up visit, unless approved by the investigator.

EXCLUSION CRITERIA:

1. Presence of self-reported or medically documented significant medical condition including but not limited to:

   1. Chronic pulmonary disease (e.g., asthma, emphysema).
   2. Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
   3. Chronic medical conditions requiring close medical follow-up or hospitalization during the past 5 years (e.g., insulin dependent diabetes mellitus, renal dysfunction, hemoglobinopathies).
   4. Immunosuppression or ongoing malignancy.
   5. Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
   6. Postinfectious or postvaccine neurological sequelae.
   7. Hyperlipidemia requiring medical therapy per current American College of Cardiology (ACC) and American Heart Association (AHA) guidelines published in 2013.
2. Have close or household (i.e., share the same apartment or house) high-risk contacts including but not limited to:

   1. Persons greater than or equal to 65 years of age.
   2. Children less than or equal to 5 years of age.
   3. Residents of nursing homes.
   4. Persons of any age with significant chronic medical conditions such as:

      * Chronic pulmonary disease (e.g., severe asthma, COPD).
      * Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
      * Contacts who required medical follow-up or hospitalization during the past 5 years because of chronic metabolic disease (e.g., insulin dependent diabetes mellitus, renal dysfunction, hemoglobinopathies).
      * Immunosuppression or cancer.
      * Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
      * Individuals who are receiving long-term aspirin therapy.
      * Women who are pregnant or who are trying to become pregnant.
3. Positive serology for hepatitis C virus antibody or hepatitis B surface antigen.
4. Individual with body mass index (BMI) greater than or equal to 18 and greater than or equal to 35 or weight > 114kg.
5. Acute illness within 7 days of admission and inoculation with the challenge virus (Day -1).
6. Complete blood count (CBC) with differential outside of the NIH Department of Laboratory Medicine (DLM) normal reference range and deemed clinically significant by the PI.
7. Chemistries in the acute care, mineral, and/or hepatic panels, and/or any of the following: lactate dehydrogenase, uric acid, creatine kinase, and total protein outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
8. Amylase or Lipase outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
9. Urinalysis outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
10. Clinically significant abnormality as deemed by the PI on electrocardiogram.
11. Clinically significant abnormality as deemed by the PI on echocardiographic (ECHO) testing.
12. Clinically significant abnormality as deemed by the PI on the Pulmonary Function Test (PFT).
13. Known allergy to treatments for influenza (including but not limited to oseltamivir, nonsteroidals).
14. Known allergy to 2 or more classes of antibiotics (e.g., penicillins, cephalosporins, fluoroquinolones, or glycopeptides).
15. Receipt of blood or blood products (including immunoglobulins) within 3 months prior to enrollment.
16. Receipt of any unlicensed drug within 3 months or 5.5 half-lives (whichever is greater) prior to enrollment.
17. Receipt of any non-influenza-related unlicensed vaccine within 6 months prior to enrollment.
18. Self-reported or known history of current alcoholism or drug abuse, or positive urine/serum test for drugs of abuse and/or ethanol (i.e., amphetamines, cocaine, benzodiazepines, opiates, or metabolites, but not tetrahydrocannabinol (THC) or metabolites).
19. Self-reported or known history of psychiatric or psychological issues deemed by the PI to be a contraindication to protocol participation.

19. Known close contact with anyone known to have influenza in the past 7 days.

21. Known or suspected hypersensitivity to CR6261 or its excipients (sucrose, L-histidine, L-histidine monohydrochloride, polysorbate 20).

22. History of a previous severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis.

23. Drinks more than 1200 mL (or 5 cups of 240 mL per cup) of tea/coffee/cocoa/cola or other caffeinated beverage per day more than 1 day per week in the 2 weeks before screening.

24. Any condition or event that, in the judgment of the PI, is a contraindication to protocol participation or impairs the volunteer s ability to give informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2015-02-25; Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Han A, Czajkowski L, Rosas LA, Cervantes-Medina A, Xiao Y, Gouzoulis M, Lumbard K, Hunsberger S, Reed S, Athota R, Baus HA, Lwin A, Sadoff J, Taubenberger JK, Memoli MJ. Safety and Efficacy of CR6261 in an Influenza A H1N1 Healthy Human Challenge Model. Clin Infect Dis. 2021 Dec 6;73(11):e4260-e4268. doi: 10.1093/cid/ciaa1725. PMID 33211860

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 104 participants signed consent and were enrolled on the protocol. 91 participants were inoculated and randomized. 13 participants did not meet criteria for influenza challenge at Day 0.
Groups:
- Placebo Comparator: Placebo, 5% dextrose (D-glucose) water
Period: Overall Study
Arm/Group | CR6261 | Placebo Comparator
Started | 49 | 42
Completed | 49 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CR6261 | Placebo Comparator | Total
Number analyzed (Participants) | 49 | 42 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 48 | 42 | 90
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 39
  Male | 32 | 20 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 40 | 34 | 74
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 13 | 34
  White | 20 | 22 | 42
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Viral Shedding
Description: Area under the curve (AUC) calculated from quantitative real-time RT-PCR for influenza A taken from 3 time per day nasal swab collection.
Time Frame: 3 times a day for 10 days
Population: All participants who were challenged with H1N1 and received CR6261
Measure: Median (Inter-Quartile Range); unit: ViralLoad(log(copies/ml))per time(hours)
Arm/Group | CR6261 | Placebo Comparator
Number analyzed (Participants) | 49 | 42
ViralLoad(log(copies/ml))per time(hours) | 48.56 [8.00 to 209.68] | 25.53 [5.00 to 159.78]
Statistical Analysis 1: Comparison: CR6261 vs Placebo Comparator; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Confirmed Influenza Infection
Description: Percentage of participants who experienced either viral shedding or symptoms + a four fold rise in convalescent HAI titer.
Time Frame: Evaluated daily for 10 days + 8 weeks convalescent follow up
Population: All participants who were challenged with H1N1 and received CR6261
Measure: Number; unit: percentage of participants
Arm/Group | CR6261 | Placebo Comparator
Number analyzed (Participants) | 49 | 42
percentage of participants | 73 | 88
Statistical Analysis 1: Comparison: CR6261 vs Placebo Comparator; Test type: Superiority; p = 0.114, Fisher Exact

3. Secondary Outcome: Days of Shedding
Description: Duration in days viral shedding was detected after influenza challenge
Time Frame: Evaluated for up to 2 months
Population: All participants who were challenged with H1N1 and received CR6261
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CR6261 | Placebo Comparator
Number analyzed (Participants) | 49 | 42
Days | 2 [1 to 4] | 2.5 [1 to 5]
Statistical Analysis 1: Comparison: CR6261 vs Placebo Comparator; Test type: Superiority; p = 0.4989, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Days of Symptoms
Description: Duration in days symptoms were experienced after influenza challenge
Time Frame: Evaluated for up to 2 months
Population: All participants who were challenged with H1N1 and received CR6261
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CR6261 | Placebo Comparator
Number analyzed (Participants) | 49 | 42
Days | 5 [3 to 7] | 6 [5 to 7]
Statistical Analysis 1: Comparison: CR6261 vs Placebo Comparator; Test type: Superiority; p = 0.1412, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Mild to Moderate Influenza Disease
Description: Percentage of participants who experienced influenza symptoms and shedding
Time Frame: Evaluated daily for 10 days
Population: All participants who were challenged with H1N1 and received CR6261
Measure: Number; unit: Percentage of participants
Arm/Group | CR6261 | Placebo Comparator
Number analyzed (Participants) | 49 | 42
Percentage of participants | 53 | 69
Statistical Analysis 1: Comparison: CR6261 vs Placebo Comparator; Test type: Superiority; p = 0.137, Fisher Exact

6. Secondary Outcome: Number of Symptoms
Description: Number of unique influenza symptoms experienced after influenza challenge
Time Frame: Evaluated for up to 2 months
Population: All participants who were challenged with H1N1 and received CR6261
Measure: Median (95% Confidence Interval); unit: Symptoms
Arm/Group | CR6261 | Placebo Comparator
Number analyzed (Participants) | 49 | 42
Symptoms | 3 [2 to 5] | 4 [3 to 5]
Statistical Analysis 1: Comparison: CR6261 vs Placebo Comparator; Test type: Superiority; p = 0.2445, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Symptoms
Description: Percentage of participants who experienced influenza symptoms
Time Frame: Evaluated daily for 10 days
Population: All participants who were challenged with H1N1 and received CR6261
Measure: Number; unit: Percentage of participants
Arm/Group | CR6261 | Placebo Comparator
Number analyzed (Participants) | 49 | 42
Percentage of participants | 76 | 93
Statistical Analysis 1: Comparison: CR6261 vs Placebo Comparator; Test type: Superiority; p = 0.045, Fisher Exact

8. Secondary Outcome: Total FLUPRO Score
Description: Objective symptoms score from patient directed FLUPRO questionnaire (inFLUenza Patient-Reported Outcome dairy) . The FLUPRO questionnaire uses a 5-point ordinal scale, with higher scores indicating a more frequent sign or symptom. Total scores can range from 0 (symptom free) to 4 (maximum severity of symptoms). Daily scores (Day 0 - Day 8) are averaged to calculate a total score for each participant, then calculated the median total FLUPRO score for each arm.
Time Frame: Evaluated from day 0 to day 8
Population: All participants who were challenged with H1N1 and received CR6261
Measure: Median (95% Confidence Interval); unit: Scores on a scale
Arm/Group | CR6261 | Placebo Comparator
Number analyzed (Participants) | 49 | 42
Scores on a scale | 0.038 [0.0125 to 0.08438] | 0.057 [0.04063 to 0.08438]
Statistical Analysis 1: Comparison: CR6261 vs Placebo Comparator; Test type: Superiority; p = 0.230, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Viral Shedding
Description: Percentage of participants who experienced influenza viral shedding
Time Frame: Evaluated daily for 10 days
Population: All participants who were challenged with H1N1 and received CR6261
Measure: Number; unit: Percentage of participants
Arm/Group | CR6261 | Placebo Comparator
Number analyzed (Participants) | 49 | 42
Percentage of participants | 67 | 74
Statistical Analysis 1: Comparison: CR6261 vs Placebo Comparator; Test type: Superiority; p = 0.646, Fisher Exact

ADVERSE EVENTS:
Time Frame: 70 days
Arm/Group | CR6261 | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/42
Other Adverse Events (participants affected / at risk) | 48/49 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CR6261 (N=49) | Placebo Comparator (N=42)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CR6261 (N=49) | Placebo Comparator (N=42)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 5 | 2
Tachycardia (Cardiac disorders) | 3 | 6
Ear discomfort (Ear and labyrinth disorders) | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 10 | 4
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 7 | 7
Oral pain (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3
Asthenia (General disorders) | 2 | 0
Chills (General disorders) | 4 | 9
Fatigue (General disorders) | 21 | 18
Non-cardiac chest pain (General disorders) | 6 | 5
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 8 | 3
Acarodermatitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 8 | 7
Hordeolum (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 31 | 31
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 4 | 3
Alanine aminotransferase increased (Investigations) | 11 | 3
Amylase increased (Investigations) | 12 | 10
Aspartate aminotransferase increased (Investigations) | 7 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 4
Blood calcium decreased (Investigations) | 1 | 0
Blood creatine phosphokinase (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 11 | 3
Blood glucose increased (Investigations) | 3 | 1
Blood phosphorus decreased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 3 | 3
Blood sodium increased (Investigations) | 3 | 2
Blood urea increased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 24 | 24
Lipase increased (Investigations) | 10 | 4
Lymphocyte count decreased (Investigations) | 3 | 7
Neutrophil count decreased (Investigations) | 16 | 11
Oxygen saturation abnormal (Investigations) | 4 | 5
Platelet count decreased (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 4 | 4
White blood cell count increased (Investigations) | 1 | 1
White blood cells urine positive (Investigations) | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 10 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Disturbance in attention (Nervous system disorders) | 2 | 2
Dizziness (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 25 | 24
Mental impairment (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 2
Bradyphrenia (Psychiatric disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 8 | 8
Nightmare (Psychiatric disorders) | 4 | 3
Haematuria (Renal and urinary disorders) | 4 | 5
Proteinuria (Renal and urinary disorders) | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 | 23
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 22 | 22
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 7
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Diastolic hypertension (Vascular disorders) | 4 | 2
Flushing (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 6 | 2
Systolic hypertension (Vascular disorders) | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT02371668/Prot_SAP_000.pdf